CLINICAL TRIAL: NCT01623102
Title: An Open-label Randomized Phase II Trial of Gemcitabine and Cisplatin With or Without Bevacizumab in EGFR Wild-type Non-squamous Non-small-cell Lung Cancer Patients
Brief Title: Cisplatin and Gemcitabine With or Without Bevacizumab in EGFR Wild-type Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Juan Li, MD, attending physician, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJP001
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: Bevacizumab; gemcitabine; cisplatin; EGFR wild-type
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: bevacizumab plus chemotherapy (Experimental): Patients in the experimental arm receive cisplatin and gemcitabine combination with Bevacizumab. GP chemotherapy (gemcitabine 1250mg/m2 IV D1 and D8 plus cisplatin 75mg/m2 IV D1, every 21-day cycle) plus bevacizumab (7.5 mg/kg IV on D1 of every 21-day cycle).
  Interventions: Drug: cisplatin and gemcitabine combination with Bevacizumab
- Arm II: chemotherapy (Active Comparator): Patients receive gemcitabine combined with cisplatin chemotherapy((gemcitabine 1250mg/m2 IV D1 and D8 plus cisplatin 75mg/m2 IV D1, every 21-day cycle) ) every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine combined with cisplatin chemotherapy

INTERVENTIONS:
Drug: cisplatin and gemcitabine combination with Bevacizumab — Patients receive gemcitabine and cisplatin chemotherapy combined with Bevacizumab every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Gemcitabine 1250mg/m2 d1, d8, cisplatin 75mg/m2 d1, Bevacizumab 7.5 mg / kg every 21 days.
  Other Names: AVASTIN
  Arms: Arm I: bevacizumab plus chemotherapy
Drug: Gemcitabine combined with cisplatin chemotherapy — Patients receive gemcitabine combined with cisplatin chemotherapy every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Gemcitabine 1250mg/m2 d1, d8, + cisplatin 75mg/m2 d1.
  Other Names: Gemzar
  Arms: Arm II: chemotherapy

SUMMARY:
Advanced non-small-cell lung cancer (NSCLC) patients without epidermal growth factor receptor (EGFR) mutations show a poor prognosis. Gemcitabine combined with cisplatin chemotherapy is an effective treatment measures for EGFR mutation-negative NSCLC patients, but the prognosis remains poor. Chemotherapy combined with targeted monoclonal antibody treatment may be better treatment options in these patients. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Bevacizumab blocks the ability of tumors to grow new blood vessels and spread. It is not yet known whether cisplatin and gemcitabine is more effective when given alone or with bevacizumab. This randomized trial studies how well giving cisplatin and gemcitabine alone or in combination with Bevacizumab (Avastin) works in treating patients with stage IIIB/IV non-squamous NSCLC without EGFR mutations.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer morbidity and mortality worldwide. The majority of lung cancer is nonsquamous NSCLC. EGFR tyrosine kinase inhibitors (EGFR-TKI) is a effective first-line treatment for EGFR mutations non-squamous NSCLC treatment. But those patients without epidermal growth factor receptor (EGFR) mutations show a poorer prognosis. Gemcitabine combined with cisplatin chemotherapy is an effective treatment measures for EGFR mutation-negative NSCLC patients, but the prognosis remains poor. Chemotherapy combined with targeted monoclonal antibody treatment may be better treatment options in these patients. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Bevacizumab blocks the ability of tumors to grow new blood vessels and spread. This randomized trial studies how well giving cisplatin and gemcitabine alone or in combination with Bevacizumab (Avastin) works in treating patients with stage IIIB/IV non-squamous NSCLC without EGFR mutations. Accordingly, we have come to a scientific hypothesis that cisplatin and gemcitabine combination with Bevacizumab might be a better treatment strategy for stage IIIB/IV non-squamous NSCLC patients with EGFR wild-type. It can improve the PFS of stage IIIB/IV non-squamous NSCLC patients with EGFR wild-type. The primary endpoint is disease-free time to progression (PFS). The secondary study endpoint is objective response rate (ORR), disease control rate (DCR), safety and quality of life (QOL). Through this study lay the foundation for further exploration of the non-squamous NSCLC first-line treatment in patients with EGFR wild-type strategy, and guide the rational application of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of primary lung carcinoma, non-squamous histology with EGFR mutation Negative.
* Stage IIIB/IV disease according to the 7th Edition of the American Joint Committee on Cancer staging system
* Not received radiotherapy, chemotherapy or other biological treatment
* Measureable disease
* Life expectancy of >= 12 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 2, 500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN in patients without liver or bone metastases; < 5 x ULN in patients with liver or bone metastases
* Cockcroft-Gault calculated creatinine clearance of >= 45 ml/min or creatinine =< 1.5 x ULN
* Prothrombin time (PT) =< 1.5 x ULN
* Partial thromboplastin time (PTT) =< ULN
* Urine dipstick proteinuria < 2+ * Note: Patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours
* Negative pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Sichuan cancer hospital for follow-up
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Prior chemotherapy or treatment for metastatic non-small cell lung cancer
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive, per MD discretion
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to randomization; EXCEPTIONS: Non melanotic skin cancer or carcinoma-in-situ of the cervix
* History of myocardial infarction or other evidence of arterial thrombotic disease (angina)
* History of cerebral vascular accident (CVA) or transient ischemic attack (TIA) =< 6 months prior to randomization
* Ongoing or active infection, symptomatic congestive heart failure , cardiac arrhythmia, psychiatric illness/social situations, or any other medical condition that would limit compliance with study requirements
* History of bleeding diathesis or coagulopathy
* Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications)
* Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury =< 28 days or core biopsy =< 7 days prior to randomization
* History of abdominal fistula, gastrointestinal perforation, or intrabdominal abscess =< 6 months prior to randomization
* History of hemoptysis >= grade 2 (defined as bright red blood of at least 2.5 mL) =< 3 months prior to randomization
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
disease-free time to progression | 6 week

SECONDARY OUTCOMES:
quality of life | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: juan li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China